CLINICAL TRIAL: NCT00831025
Title: Multicenter, Randomised, Double-blind Placebo-controlled, Subcutaneous Immunotherapy Clinical Trial With Depigmented and Polymerized Allergen Extract of Olea Europaea Pollen in Patients With Hypersensitivity to Olea Pollen
Brief Title: Subcutaneous Immunotherapy Treatment for Patients With Hypersensitivity to Olea Europaea Pollen
Acronym: OLEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6018-PG-PSC-148; 2006-005727-41 (EudraCT Number)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Rhinitis or Rhinoconjunctivitis With or Without Asthma Induced by Hypersensitivity to Olea Europea Pollen
Keywords: Immunotherapy; Allergoid; Depigmented; Polymerized; Allergen-extract; Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis | interventions — Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Depigmented and polymerized allergen extract of Olea europaea pollen for subcutaneous injection.
  Interventions: Biological: Immunotherapy with modified extract of Olea europaea pollen
- 2 (Placebo Comparator): Placebo for subcutaneous injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Immunotherapy with modified extract of Olea europaea pollen — Subcutaneous immunotherapy with modified extract of Olea europaea. A subcutaneous monthly treatment.
  Arms: 1
Biological: Placebo — Placebo for subcutaneous monthly administration
  Arms: 2

SUMMARY:
The objective of this trial is to assess the clinical efficacy of a modified allergen extract of Olea europaea pollen in the treatment of patients affected by allergic rhinitis/rhinoconjunctivitis (with or without episodic asthma) induced by hypersensitivity to olea europaea pollen, evaluating the Score regarding Symptoms and consumption of the medication.

DETAILED DESCRIPTION:
Immunotherapy is a specific treatment for allergic diseases. Unlike conventional pharmacological treatment, immunotherapy is the only treatment that could modify the natural course of allergic disease. This is a prospective double-blind placebo-controlled study with two arms of treatment: placebo and active.

ELIGIBILITY:
Inclusion Criteria:

* Prior to study specific examinations the patient and if applicable both legal guardians has to give his/her written informed consent
* Patients of both gender aged from 18 and 55 years
* Patient's perception of disease activity of at least 30 mm on a 100 mm visual analogue scale (VAS)
* FEV1 greater or equal than 80% of the expected value, and if not, improvement of FEV1 greater than 12% after bronchodilation
* Patients have to suffer from allergic complaints (rhinitis and/or rhinoconjunctivitis with or without mild intermittent allergic asthma) caused by clinical sensitization against Olea europaea pollen. The IgE mediated sensitization has to be verified by:
* Suggestive medical history
* Specific IgE against Olea europaea pollen CAP RAST ≥0.7Ku/l
* Positive skin prick test (SPT) to grass Olea pollen resulting in a wheal diameter of at least 3 mm.

Exclusion Criteria

* History of significant clinical manifestations of allergy as a result of sensitization against weed pollen allergens and perennial (e.g. house dust mite.
* Participation in an immunotherapy with comparable extracts within the last five years.
* Treatment with β-blocker
* Any disease which prohibits the use of adrenaline (e.g. hyperthyroidism)
* Cardiovascular insufficiency or any severe or unstable pulmonary, or endocrine disease; clinically significant renal or hepatic disease or dysfunction; hematologic disorder; any other clinically significant medical condition that could increase the risk to the study participant
* Immunopathological diseases
* Patients who are expected to be non-compliant and/or not co-operative
* Women, where pregnancy is defined as the state of a female after conception and until the termination of gestation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Symptoms and medication score | 2 years

SECONDARY OUTCOMES:
Dose-response skin prick-test | 2 years
Medication score | 2 years
Rhinoconjunctivitis quality of life questionnaire | 2 years
Visual Analog Scales (VAS) | 2 years
Serology | 2 years
Symptoms score | 2 years
Exhaled nitric oxide | 2 years
Adverse event | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Guardia, MD, Principal Investigator
Locations (7):
- Spain (7):
  - Hospital El Tomillar, Dos Hermanas, Sevilla
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Virgen Del Rocio, Seville
  - Clínica Santa Isabel, Seville
  - Hospital Virgen Macarena, Seville